CLINICAL TRIAL: NCT02003534
Title: A Study of 0.15% Brimonidine Tartrate in Patients With Primary Open Angle Glaucoma and Ocular Hypertension
Acronym: APOTUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN-BRI-1002
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-06

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.15% Brimonidine Tartrate (Experimental): 0.15% Brimonidine Tartrate (Alphagan® P) 1 drop in the affected eye 3 times daily for 3 months.
  Interventions: Drug: 0.15% Brimonidine Tartrate

INTERVENTIONS:
Drug: 0.15% Brimonidine Tartrate — 0.15% Brimonidine Tartrate (Alphagan® P) 1 drop in the affected eye 3 times daily for 3 months.
  Other Names: Alphagan® P

SUMMARY:
This study will evaluate 0.15% brimonidine tartrate in patients with primary open angle glaucoma and ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* Used Alphagan® in previous 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2010-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Shanghai, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.15% Brimonidine Tartrate
Started | 376
Completed | 329
Not Completed | 47
Not completed — Lost to Follow-up | 47

BASELINE CHARACTERISTICS:
Arm/Group | 0.15% Brimonidine Tartrate
Number analyzed (Participants) | 376
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161
  Male | 215

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) in the Study Eye
Description: IOP is a measurement of the fluid pressure inside the eye. A negative number change from baseline indicates a reduction in IOP (improvement), and a positive number change from baseline indicates an increase (worsening).
Time Frame: Baseline, Month 3
Population: Intent-to-Treat: patients with baseline data and data at the indicated time point
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | 0.15% Brimonidine Tartrate
Number analyzed (Participants) | 376
Millimeters of Mercury (mmHg)
  Baseline | 25.4 (2.3)
  Change from Baseline at Month 3 (N=330) | -6.3 (3.5)

ADVERSE EVENTS:
Description: The Safety Set included all treated patients and was used to evaluate adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | 0.15% Brimonidine Tartrate
Serious Adverse Events (participants affected / at risk) | 0/372
Other Adverse Events (participants affected / at risk) | 24/372
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.15% Brimonidine Tartrate (N=372)
Conjunctiva Hyperemia (Eye disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.